CLINICAL TRIAL: NCT07351201
Title: The Effect of Head and Neck Positioning on Lung Sliding: A Bedside Comparison at 0°, 20°, and 40° in Healthy Volunteer
Brief Title: Effect of Head and Neck Positioning on Lung Sliding in Healthy Volunteers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, İLKER ŞİRİN, Specialist Physician, Ankara Etlik City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AEŞH-EK-2025-305
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Ultrasonography; Lung; Pleura; Respiratory Mechanics; Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Head-of-Bed Position Assessment (0°, 20°, 40°) (Other): Participants in this single-arm study will undergo lung ultrasound assessments during a single study visit. Each participant will be positioned sequentially at three different head-of-bed angles: zero degrees (supine), twenty degrees, and forty degrees. At each position, lung sliding movement will be evaluated using bedside lung ultrasonography with a high-frequency linear probe.
  Measurements will be obtained from four predefined anatomical regions: right apical, right basal, left apical, and left basal lung areas. Lung sliding will be quantitatively assessed using M-mode imaging by measuring pleural line displacement.
  Interventions: Procedure: Head-of-Bed Elevation

INTERVENTIONS:
Procedure: Head-of-Bed Elevation — Controlled positioning of the participant with the head of the bed at zero, twenty, and forty degrees. At each position, lung sliding movement will be assessed using bedside lung ultrasound with a high-frequency linear probe.

SUMMARY:
The goal of this clinical study is to learn how different head-of-bed positions affect lung movement during breathing in healthy adults. Researchers want to understand whether raising the head of the bed changes how the lungs move, which may help guide patient positioning in emergency and intensive care settings.

The main questions this study aims to answer are:

Does lung movement change when the head of the bed is positioned at zero, twenty, or forty degrees?

Are there differences in lung movement between the right and left lungs?

Are there differences between the upper (apical) and lower (basal) parts of the lungs?

Participants will be healthy adult volunteers between eighteen and sixty years of age. Each participant will lie on a bed in three different positions: flat, with the head raised to twenty degrees, and with the head raised to forty degrees.

During each position, researchers will use bedside lung ultrasound, a painless and non-invasive imaging method, to measure lung movement at four areas of the chest. No medications, injections, or invasive procedures will be used.

This study may help health care providers better understand how body position affects breathing and support safer and more effective positioning of patients with breathing problems.

DETAILED DESCRIPTION:
This is a prospective, low-risk, non-drug interventional clinical study designed to evaluate the effect of head-of-bed elevation on lung sliding movement in healthy adult volunteers. Lung sliding is a dynamic ultrasound finding that reflects the movement between the visceral and parietal pleura during respiration and provides information about lung aeration and respiratory mechanics.

The primary objective of the study is to quantitatively assess changes in lung sliding amplitude across three standardized head-of-bed positions: zero degrees (supine), twenty degrees, and forty degrees. Measurements will be obtained using bedside lung ultrasonography at four predefined anatomical locations: right apical, right basal, left apical, and left basal lung regions.

Secondary objectives include evaluating potential differences in lung sliding between the right and left lungs, comparing apical and basal lung regions, and assessing whether positional changes have region-specific effects on lung movement.

The study population will consist of thirty-one healthy adult volunteers aged eighteen to sixty years. Individuals with known respiratory disease, significant cardiopulmonary conditions, pregnancy, prior thoracic surgery, or inability to tolerate position changes will be excluded. All participants will provide written informed consent prior to enrollment.

Each participant will undergo lung ultrasound measurements in all three positions in a repeated-measures design. Lung sliding will be recorded using high-frequency linear ultrasound probes. Quantitative assessment will be performed using M-mode imaging, measuring pleural line displacement in millimeters. Mean values will be calculated for each position and anatomical region.

No investigational drugs, medical devices, or invasive procedures will be used. The only intervention is controlled head-of-bed positioning. The study is considered minimal risk. Potential discomfort related to short-term position changes, such as mild dizziness or transient shortness of breath, will be monitored, and measurements will be discontinued if symptoms occur.

Data will be analyzed using repeated measures statistical methods to compare lung sliding values across positions and regions. The findings are expected to improve understanding of the positional sensitivity of lung ultrasound measurements and may contribute to evidence-based recommendations for patient positioning in emergency and critical care settings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers aged eighteen to sixty years.
* No history of acute or chronic respiratory disease.
* Body mass index between eighteen point five and twenty-nine point nine kilograms per square meter.
* Ability to understand the study procedures and provide written informed consent.
* No skin lesions or wounds at the chest wall that would interfere with lung ultrasound examination.

Exclusion Criteria:

* History of respiratory system diseases, including asthma, chronic obstructive pulmonary disease, bronchiectasis, pneumonia, or tuberculosis.
* Presence of chest wall deformities (such as kyphoscoliosis or pectus deformities) or history of thoracic surgery.
* Inability to tolerate position changes during the study, including development of dizziness, syncope, or shortness of breath.
* Pregnancy or breastfeeding.
* Known significant cardiac, neurological, or metabolic disease.
* Known allergy to ultrasound gel or latex.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in Lung Sliding Amplitude Across Different Head-of-Bed Positions | Periprocedural (during a single study visit)
  Lung sliding amplitude will be quantitatively measured using bedside lung ultrasonography in healthy adult participants. Measurements will be obtained at four predefined anatomical regions (right apical, right basal, left apical, and left basal lung areas) while participants are positioned sequentially at three head-of-bed angles: zero degrees, twenty degrees, and forty degrees. Lung sliding amplitude will be assessed using M-mode imaging by measuring pleural line displacement in millimeters. Mean values for each position will be calculated and compared to evaluate the effect of head-of-bed elevation on lung sliding movement.

SECONDARY OUTCOMES:
Difference in Lung Sliding Amplitude Between Right and Left Lungs | Periprocedural (during a single study visit)
  Lung sliding amplitude values obtained from the right and left lungs will be compared to assess side-related differences in lung movement. Measurements will be performed at both apical and basal regions of each lung using bedside lung ultrasonography while participants are positioned at three different head-of-bed angles (zero, twenty, and forty degrees). This analysis will evaluate whether lung sliding differs between the right and left lungs under different positional conditions.

CONTACTS AND LOCATIONS:
Overall Officials: İLKER ŞİRİN, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study involves a small sample of healthy volunteers and collects detailed physiological measurements that could increase the risk of re-identification, even after de-identification. The study protocol and informed consent do not include provisions for public sharing of individual-level data. Only aggregated and anonymized results will be reported.

REFERENCES:
- [Background] Nelson DM, Johnson RD, Smith SD, Anteby EY, Sadovsky Y. Hypoxia limits differentiation and up-regulates expression and activity of prostaglandin H synthase 2 in cultured trophoblast from term human placenta. Am J Obstet Gynecol. 1999 Apr;180(4):896-902. doi: 10.1016/s0002-9378(99)70661-7. PMID 10203658
- [Background] Sirin I, Erdem AB, Uysal SB, Gedikaslan S. The Effect of Tidal Volumes of Mechanically Ventilated Patients on Lung Sliding Amplitude in Point-Of-Care Lung Ultrasound. J Clin Ultrasound. 2025 Jun;53(5):989-996. doi: 10.1002/jcu.23968. Epub 2025 Mar 17. PMID 40098375